CLINICAL TRIAL: NCT03461588
Title: Prospective Assessment of Radiation-induced Heart Injury in Left-sided Breast Cancer Treated With Breast Conserving Surgery Followed by Radiotherapy With Free-breathing or Deep Inspiration Breath-hold (DIBH) Technique
Brief Title: Prospective Assessment of Radiation-induced Heart Injury in Left-sided Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shu lian Wang (Unknown)
Responsible Party: Sponsor-Investigator, Shu lian Wang, professor of medicine, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2016A09
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Breast Neoplasms; Heart Injuries; Radiation Toxicity
MeSH Terms: conditions — Breast Neoplasms; Heart Injuries; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Free-breathing (Active Comparator): standard treatment
  Interventions: Radiation: free-breathing
- Deep inspiratory breath-holding (Experimental): new technique
  Interventions: Radiation: deep inspiratory breath-holding

INTERVENTIONS:
Radiation: free-breathing — patients are irradiated to whole breast +- regional nodal areas with free-breathing technique after breast conserving surgery
  Arms: Free-breathing
Radiation: deep inspiratory breath-holding — patients are irradiated to whole breast +- regional nodal areas with deep inspiratory breast-holding technique after breast conserving surgery
  Arms: Deep inspiratory breath-holding

SUMMARY:
This study is to prospectively investigate the cardiac dose-sparing effect and clinical benefit of deep inspiration breath-hold (DIBH) technique. Patients with left-sided breast cancer treated with breast conserving surgery followed by radiotherapy is enrolled. Radiotherapy is delivered with either free-breathing or deep inspiration breath-hold (DIBH) technique. The cardiac dose parameters and cardiac toxicity are prospective evaluated, and the dose-effect relationship is analyzed.

DETAILED DESCRIPTION:
Patients with left-sided breast cancer treated with breast conserving surgery are prospectively enrolled. Two types of radiation treatment are delivered based on attending physician's preferences: radiation to whole breast +- regional nodal areas with free-breathing technique, or with deep inspiration breath-hold (DIBH) technique. The cardiac dose parameters including heart dose and the dose to left anterior coronary artery are assessed, and the cardiac toxicities regularly assessed with cardiac enzymes,electrocardiogram(ECG) and normal gated single-photon emission computed tomography-myocardial perfusion imaging before, during and after radiation.The dose-effect relationship of heart injuries is analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Left-sided breast cancer
2. Underwent breast conserving surgery
3. Planned for postoperative whole breast +- regional nodal radiotherapy
4. No basic heart disease

Exclusion Criteria:

1. Abnormal cardiac baseline examination
2. History of chest radiation
3. Can not tolerate deep inspiratory breath-holding

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female only
Enrollment: 140 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related cardiac adverse events as assessed by CTCAE v4.0 | up to 2 years
  The cardiac adverse events are regularly assessed with cardiac symptoms,cardiac enzymes(TnT，BNP),electrocardiogram(ECG) and normal gated single-photon emission computed tomography-myocardial perfusion imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Shulian Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Cancer Hosptical, Chinese Academy of Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No